CLINICAL TRIAL: NCT06519227
Title: Translation and Validation of Urdu Version of the Rivermead Mobility Index in Stroke Survivors
Brief Title: Translation and Validation of Rivermead Mobility Index in Urdu
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/31
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Stroke Patients
Keywords: stroke, sub-acute stroke, translation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rivermead Mobility Index (RMI) is an internationally used tool to assess mobility for both research and clinical practice in stroke survivors. This tool had previously been translated into many languages. However, the Urdu version of RMI is not available yet.

The purpose of this study was to translate the RMI into Urdu (RMI-U) and to evaluate the validity and reliability of the translated version among Urdu-speaking stroke survivors in Pakistan. A standardized stepwise forward-backward translation procedure following international guidelines, was used to translate RMI into Urdu. The RMI-U pre-final version underwent thorough psychometric testing. Content validity was evaluated by measuring content validity indices (CVIs). The test-retest reliability of final version was then evaluated among 150 stroke survivors after a one-week interval. Furthermore, internal consistency was measured by Cronbach's alpha and construct validity by exploring factor analysis using the principle of component extraction and a Varimax rotation.

DETAILED DESCRIPTION:
Stroke is the second most common cause of death and the third most common cause of disability in adults worldwide including in Asia. Stroke survivors experience varying degrees of sensory-motor impairments including lack of mobility, reduced functional activity, and poor coordination and balance either due to muscular weakness or spasticity. Mobility is adversely affected after stroke, as patients may face many problems in moving and getting around (walking, stair climbing, etc) .

In stroke rehabilitation, it is recommended to evaluate mobility deficits using standardized tools. RMI is a valid and reliable tool, used internationally for its appropriate psychometric properties. It is used in stroke patients as a marker of mobility, which assesses balance, mobility, transfer, and gait in stroke survivors. Originally it was developed in 1991 in English language. and translated into different languages for its feasibility and responsiveness such as German, Italian, Turkish, and Brazilian, Dutch, and Danish.

Stroke is a major public health concern in developing countries of South Asia including Pakistan. The estimated incidence rate of stroke in Pakistan is 250/100,000 annually. Currently, English RMI is used for the clinical evaluation of mobility in stroke patients. Whereas Urdu is the public language of Pakistani people and most of the patients suffering from stroke belong to rural areas of Pakistan, where the literacy rate is low, and a small proportion of the population can read and understand English. Due to the language barrier and moderate pace of education, it's difficult to them to understand English language. Therefore, its Urdu translation was needed. As per knowledge of the author no Urdu version of RMI is available yet. So, this study aimed to develop Urdu version RMI-U and to test the validity and reliability of the translated version in stroke patients. So that in future it can be easily implemented throughout the Pakistani healthcare system and its utility in public and private healthcare setup could increase.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic stroke; ischemic or hemorrhagic,
* Aged between 40 to 80 years who visited the respective rehabilitation center during the study time
* Those who could read and understand Urdu.

Exclusion Criteria

Ages: 45 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Whereas those with cognitive impairment, Broca aphasia Wernicke s aphasia or with other neurological disorder e.g. previous cranial traumatic injuries tumors
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Rivermead Mobility Index | 2nd day
  mobility assessment

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, phD*, Principal Investigator — Riphah International University
Locations (1):
- Binash Afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossier P, Wade DT. Validity and reliability comparison of 4 mobility measures in patients presenting with neurologic impairment. Arch Phys Med Rehabil. 2001 Jan;82(1):9-13. doi: 10.1053/apmr.2001.9396. PMID 11239279
- [Background] Franchignoni F, Tesio L, Benevolo E, Ottonello M. Psychometric properties of the Rivermead Mobility Index in Italian stroke rehabilitation inpatients. Clin Rehabil. 2003 May;17(3):273-82. doi: 10.1191/0269215503cr608oa. PMID 12735534
- [Background] Pavan K, da Cruz LC, Nunes MF, Menezes LG, Marangoni BE. Cross-cultural adaptation and validation of the Rivermead Mobility Index in stroke patients within the brazilian cultural and language context. Arq Neuropsiquiatr. 2010 Feb;68(1):52-5. doi: 10.1590/s0004-282x2010000100012. PMID 20339653
- [Background] Roorda LD, Green J, De Kluis KR, Molenaar IW, Bagley P, Smith J, Geurts AC. Excellent cross-cultural validity, intra-test reliability and construct validity of the Dutch Rivermead Mobility Index in patients after stroke undergoing rehabilitation. J Rehabil Med. 2008 Oct;40(9):727-32. doi: 10.2340/16501977-0249. PMID 18843424
- [Background] Steen Krawcyk R, Hagell P, Sjodahl Hammarlund C. Danish translation and psychometric testing of the Rivermead Mobility Index. Acta Neurol Scand. 2013 Oct;128(4):e20-5. doi: 10.1111/ane.12144. Epub 2013 Jun 13. PMID 23758575